CLINICAL TRIAL: NCT02011165
Title: An Objective Evaluation of Postoperative Positioning in Macular Hole Surgery
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REK2013/781
Record Dates: First submitted 2013-12-04; First posted 2013-12-13 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Macular Hole
Keywords: Macular hole; Vitrectomy; Gas tamponade; Vitreomacular traction in danger of macular hole formation; Epiretinal membrane in danger of macular hole formation
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tennis ball: Night with tennis ball fastened in the back of the night shirt. A positioning measuring device mounted.
  Interventions: Procedure: Positioning measuring device
- No tennis ball: Night without tennis ball fastened in the back of the night shirt. A positioning measure device mounted.
  Interventions: Procedure: Positioning measuring device

INTERVENTIONS:
Procedure: Positioning measuring device — A tennis ball in the night shirt will prevent supine position during sleep.
  Other Names: Measurement of time spent in the supine position

SUMMARY:
The macular hole formation takes place in the centre of the retina. A closure of the macular hole is believed to take place if the central retinal area is kept dry in the postoperative period. Therefore the eye is filled with a gas mix and the patients are urged to avoid the supine position in the first postoperative days. The investigators use the "tennis ball technique" where a tennis ball is fastened in the back of the night shirt in order to help patients compliance in avoiding the supine sleeping position. The investigators have developed a positioning measuring device which can measure the extent of supine positioning time. Patients are to sleep two nights with the positioning measuring device, one night with a tennis ball in the back of the night shirt and one night without. Hereby the investigators search new knowledge concerning patients compliance and verification of the "tennis ball technique".

ELIGIBILITY:
Inclusion Criteria:

* Pars plana vitrectomy for macular hole, vitreomacular traction or epiretinal membrane where intra ocular gas tamponade is used.
* Informed consent

Exclusion Criteria:

* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing pars plana vitrectomy for macular hole formation, or conditions as epiretinal menbrane or vitreomacular traction where a macular hole formation is likely.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time in supine sleeping position | Two days

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Forsaa, MD, Principal Investigator — Helse Stavanger HF
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Stavanger University Hospital, Department of Ophthalmology, Stavanger

REFERENCES:
- [Background] Forsaa VA, Raeder S, Hashemi LT, Krohn J. Short-term postoperative non-supine positioning versus strict face-down positioning in macular hole surgery. Acta Ophthalmol. 2013 Sep;91(6):547-51. doi: 10.1111/j.1755-3768.2012.02464.x. Epub 2012 Jul 25. PMID 22830524